CLINICAL TRIAL: NCT06751459
Title: Patch ECG-based REcurrEnce Monitoring After Catheter Ablation in PaTients with Atrial Fibrillation (PREEMPT-AF) : a Multicenter, Randomized Controlled, Open-label, Prospective Trial
Brief Title: Evaluation of the Effectiveness and Safety of Remote Electrocardiographic Monitoring in Patients with Atrial Fibrillation Following Ablation Therapy
Acronym: PREEMPT-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HUINNO Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PREEMPT-AF
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial fibrillation; circulatory system; EKG; remote monitoring; gateway; MEMO-Patch
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants in this clinical trial will undergo a total of three remote electrocardiographic (ECG) monitoring sessions during the study period following catheter ablation:
  1. st Monitoring: At the time of discharge after catheter ablation, remote ECG monitoring will be performed for 14 days using both the MEMO Patch 2 and MEMO Link.
  2. nd Monitoring: Approximately three months after catheter ablation, remote ECG monitoring will be performed for 14 days using only the MEMO Patch 2.
  3. rd Monitoring: Approximately one year after catheter ablation, remote ECG monitoring will again be performed for 14 days using only the MEMO Patch 2.
  Interventions: Device: MEMO Patch 2 - 1-day Monitoring; Device: MEMO Link
- Active Comparator Group (Active Comparator): Participants in this clinical trial will undergo a total of three remote electrocardiographic (ECG) monitoring sessions during the study period following catheter ablation:
  1. st Monitoring: At the time of discharge after catheter ablation, remote ECG monitoring will be conducted for 14 days using both the MEMO Patch 2 and MEMO Link.
  2. nd Monitoring: Approximately three months after catheter ablation, remote ECG monitoring will be conducted for 1 day using only the MEMO Patch 2.
  3. rd Monitoring: Approximately one year after catheter ablation, remote ECG monitoring will be conducted for 14 days using only the MEMO Patch 2.
  Interventions: Device: MEMO Patch 2 - 14-day Monitoring; Device: MEMO Link

INTERVENTIONS:
Device: MEMO Patch 2 - 14-day Monitoring — A wearable ECG monitoring device used for continuous 14-day monitoring to detect atrial arrhythmias during the second monitoring phase (at 3 months post-ablation). MEMO Patch 2 collects ECG data for remote analysis to assess early recurrence of atrial arrhythmias.
  Arms: Active Comparator Group
Device: MEMO Patch 2 - 1-day Monitoring — A wearable ECG monitoring device used for 1-day monitoring during the second monitoring phase (at 3 months post-ablation). MEMO Patch 2 collects ECG data for remote analysis to detect early recurrence of atrial arrhythmias.
  Arms: Experimental Group
Device: MEMO Link — A supplementary ECG monitoring device used alongside MEMO Patch 2 during the 1st monitoring session.

SUMMARY:
Background:

Atrial fibrillation (AF) is the most common arrhythmia, significantly contributing to complications such as stroke, heart failure, dementia, and increased mortality. Catheter ablation is widely used for treatment, but recurrence rates range from 15-50% within 12 months post-procedure. Conventional intermittent ECG monitoring lacks sufficient sensitivity to detect asymptomatic AF recurrence effectively.

Objective:

To compare the recurrence rates of atrial tachyarrhythmias between a 1-day monitoring group and a 14-day monitoring group using MEMO Patch 2 after catheter ablation in AF patients. The study also evaluates the effectiveness and safety of early recurrence detection via remote monitoring.

Study Population:

Patients diagnosed with AF and treated with catheter ablation.

Intervention:

Participants will undergo three sessions of remote ECG monitoring using MEMO Patch 2 and MEMO Link (first session only), spanning approximately one year after catheter ablation.

Hypothesis:

Long-term monitoring with MEMO Patch 2 will be more effective than 1-day monitoring in detecting the recurrence of atrial tachyarrhythmias (including AF, atrial flutter, and atrial tachycardia) following catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 19 years or older who have voluntarily provided written informed consent to participate in this clinical trial.

  2. Individuals who have been diagnosed with atrial fibrillation prior to the date of informed consent acquisition.

  3. Individuals who are scheduled to undergo catheter ablation for atrial fibrillation within three months from the date of informed consent acquisition.

Exclusion Criteria:

* 1. Individuals with a history of catheter ablation prior to obtaining informed consent.

  2. Individuals with sensitive skin, allergic skin conditions, skin cancer, rashes, or other dermatological disorders.

  3. Individuals with implanted cardiac devices, such as pacemakers, implantable defibrillators, or other implantable electronic devices.

  4. Individuals deemed by the investigator to be at an increased risk or otherwise unsuitable for participation in the clinical trial.

  5. Individuals with cognitive impairments that make it difficult to understand trial information or voluntarily make an informed decision.

  6. Pregnant or breastfeeding women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of atrial tachyarrhythmias 3 months post-catheter ablation | 3 months post-ablation
  The proportion of participants with atrial tachyarrhythmias (including atrial fibrillation, atrial flutter, or atrial tachycardia lasting 30 seconds or more) detected during ECG monitoring at 3 months after catheter ablation using the MEMO Patch 2. The primary measure focuses on comparing the detection rate between the 14-day monitoring group and the 1-day monitoring group.

SECONDARY OUTCOMES:
Risk Factors for Early and Late Recurrence of Atrial Tachyarrhythmias | 12 months post-ablation
  Identification of clinical risk factors associated with early recurrence (within 3 months) and late recurrence (beyond 3 months) of atrial tachyarrhythmias following catheter ablation, using data collected through MEMO Patch 2 monitoring.
Rate of Medical Interventions Following Catheter Ablation | 12 months post-ablation
  Proportion of participants requiring additional medical interventions such as anti-arrhythmic drug cessation, repeat ablation procedures, or unplanned clinical visits post-ablation.
Recurrence Rate of Atrial Tachyarrhythmias at 12 Months | 12 months post-ablation
  Proportion of participants experiencing atrial tachyarrhythmias (lasting 30 seconds or more) detected by MEMO Patch 2 within 12 months after catheter ablation.
Early Recurrence Rate of Atrial Tachyarrhythmias | 3 months post-ablation
  Proportion of participants with atrial tachyarrhythmias detected within 3 months post-ablation using MEMO Patch 2.
Detection Rate of Non-Atrial Tachyarrhythmias Using MEMO Patch 2 | 12 months post-ablation
  Proportion of participants with non-atrial tachyarrhythmias, such as ventricular premature contractions or supraventricular tachycardia, detected during MEMO Patch 2 monitoring.
Time to First Recurrence of Atrial Tachyarrhythmias | 12 months post-ablation
  The time interval from catheter ablation to the first detection of atrial tachyarrhythmias lasting 30 seconds or more during MEMO Patch 2 monitoring.
ECG Signal Transmission Success Rate Using MEMO Link | During all monitoring periods (up to 12 months post-ablation)
  Percentage of successfully transmitted ECG signals during the monitoring period using the MEMO Link device.
Detection Rate of Atrial Tachyarrhythmias in Daily Monitoring Reports | 30 days post-ablation (first monitoring phase)
  Proportion of participants with atrial tachyarrhythmias detected using daily ECG monitoring reports during the first monitoring phase (up to 30 days post-ablation).
Device-Related Adverse Events | During all monitoring periods (up to 12 months post-ablation)
  Rate of adverse events potentially related to the use of MEMO Patch 2 or MEMO Link during the study period, assessed through investigator reports.

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Dong-A University Hospital, Busan
  - Busan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including basic demographic data and primary research outcome data, will be shared. These data will specifically pertain to research conducted on remote monitoring and atrial fibrillation. The shared data will not contain any personal identifiers to ensure participant
  When the data are made available, a direct link to the external repository hosting the IPD will be provided in the References module of the Protocol Section on ClinicalTrials.gov.
Access Criteria: Qualified researchers may request access to the IPD by submitting a formal application. Requests must include a detailed research proposal and evidence of ethical approval. All requests will be reviewed by an independent committee to ensure appropriate and ethical use of the data. Once a suitable data-sharing platform or repository is designated, detailed instructions for access will be provided in the ClinicalTrials.gov record.